CLINICAL TRIAL: NCT06265883
Title: Lenvatinib Plus Drug-eluting Bead Transarterial Chemoembolization and Hepatic Arterial Infusion Chemotherapy Versus Lenvatinib Plus Drug-eluting Bead Transarterial Chemoembolization for Large Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis: a Multicenter Retrospective Cohort Study
Brief Title: Lenvatinib Plus DEB-TACE With/Without FOLFOX-HAIC for Large HCC With PVTT
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Zhongshan People's Hospital, Guangdong, China (Other); Affiliate Hospital of Guangdong Medical University (Unknown); Jieyang People's Hospital (Other); Huizhou Municipal Central Hospital (Other); Guangzhou Development District Hospital (Unknown); Affiliated Hospital of Nanjing University of Chinese Medicine (Other); First People's Hospital of Foshan (Other)
Responsible Party: Sponsor
Other Study IDs: MIIR-16-Retro
Record Dates: First submitted 2024-02-10; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular Carcinoma; Lenvatinib; transarterial chemoembolization; drug-eluting bead; hepatic arterial infusion chemotherapy; portal vein tumor thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Len+DEB-TACE+HAIC: Patients were treated with Len+DEB-TACE+HAIC.
  Interventions: Procedure: Len+DEB-TACE+HAIC
- Len+DEB-TACE: Patients were treated with Len+DEB-TACE.
  Interventions: Procedure: Len+DEB-TACE

INTERVENTIONS:
Procedure: Len+DEB-TACE+HAIC — Patients received TACE with drug-eluting beads and FOLFOX-HAIC. DEB-TACE and/or HAIC was repeated for viable tumors demonstrated by follow-up imaging in patients without worsening liver function or contraindications. Lenvatinib was orally administered at a dose of 12 mg/day (bodyweight 60 kg) or 8mg/day (bodyweight <60 kg). It was initiated within 7 days after the first DEB-TACE or DEB-TACE+HAIC and continued until unacceptable toxicity or disease progression occurred.
  Groups: Len+DEB-TACE+HAIC
Procedure: Len+DEB-TACE — Patients received TACE with drug-eluting beads. DEB-TACE was repeated for viable tumors demonstrated by follow-up imaging in patients without worsening liver function or contraindications. Lenvatinib was orally administered at a dose of 12 mg/day (bodyweight 60 kg) or 8mg/day (bodyweight <60 kg). It was initiated within 7 days after the first DEB-TACE or DEB-TACE+HAIC and continued until unacceptable toxicity or disease progression occurred.
  Groups: Len+DEB-TACE

SUMMARY:
This multicenter retrospective study evaluated consecutive patients with large HCC and PVTT who received lenvatinib plus DEB-TACE with/without FOLFOX-HAIC between July 2019 and June 2021. Tumor response, time to progression (TTP), overall survival (OS), and treatment-related adverse events (TRAEs) were compared between the two groups.

DETAILED DESCRIPTION:
Consecutive patients with large HCC and PVTT treated with lenvatinib plus drug-eluting bead transarterial chemoembolization (DEB-TACE) and hepatic arterial infusion chemotherapy (HAIC) with oxaliplatin, fluorouracil and leucovorin (Len+DEB-TACE+HAIC) or lenvatinib plus DEB-TACE (Len+DEB-TACE) from July 2019 to June 2021 were screened. Tumor response was evaluated according to modified Response Evaluation Criteria in Solid Tumors (mRECIST). Clinical outcomes, including tumor response, TTP, OS, and TRAEs were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of HCC
* the largest intrahepatic lesion >7 cm
* presence of major PVTT on imaging
* Eastern Cooperative Oncology Group performance status ≤1
* Child-Pugh class A/B
* adequate hematologic and organ function, with leukocyte count 3.0 109/L, neutrophil count 1.5 109/L, platelet count 75 109/L, hemoglobin 85 g/L, alanine transaminase and aspartate transaminase 5 upper limit of the normal, creatinine clearance rate 1.5 upper limit of the normal, and prothrombin time prolongation <4 s

Exclusion Criteria:

* incomplete medical records
* central nervous system involvement
* previous treatment with transarterial embolization, TACE, HAIC, radiotherapy, or systemic therapy
* history of malignancies other than HCC
* history of organ transplantation
* severe cardiac, pulmonary or renal dysfunction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with large HCC and PVTT.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | 3.5 years
  defined as the time from treatment initiation to the first occurrence of disease progression.

SECONDARY OUTCOMES:
objective response rate (ORR) | 3.5 years
  defined as the percentage of patients with complete or partial response
Disease control rate (DCR) | 3.5 years
  defined as the percentage of patients with complete or partial response, or stable disease
overall survival | 3.5 years
  defined as the time from treatment initiation until death from any reason.
treatment-related adverse events (TRAEs) | 3.5 years
  assessed based on Common Terminology Criteria for Adverse Events version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cai M, Liang L, Zhang J, Chen N, Huang W, Guo Y, Hong X, Lin L, Liu Y, Dan C, Deng H, Liu X, Zhou J, Chen Y, Chen H, Zhu K. Lenvatinib plus drug-eluting bead transarterial chemoembolization with/without hepatic arterial infusion chemotherapy for hepatocellular carcinoma larger than 7 cm with major portal vein tumor thrombosis: a multicenter retrospective cohort study. Int J Surg. 2024 Dec 1;110(12):7860-7870. doi: 10.1097/JS9.0000000000001819. PMID 38869974